CLINICAL TRIAL: NCT05762692
Title: Clinical Feasibility and Efficacy of High-flow Nasal Oxygenation During Intravenous Deep Sedation in Pediatric Dental Patients
Brief Title: High-flow Nasal Oxygenation During Deep Sedation in Pediatric Dental Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Xudong, Chief of Department of Anesthesiology, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PKUSSIRB-202283174
Record Dates: First submitted 2023-02-09; First posted 2023-03-10 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Deep Sedation; Dental Treatment; Pediatric Patients
Keywords: high-flow nasal oxygenation; dental treatment; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFNO Group (Experimental): Intra-operative oxygenation will be administered by the high-flow nasal oxygenation device. The flow rate is 2L/kg.(upper limit 30L/min)
  Interventions: Device: High-flow nasal oxygenation device

INTERVENTIONS:
Device: High-flow nasal oxygenation device — The patients included will be oxygenated by HFNO device during the operation

SUMMARY:
It is important to choose an appropriate oxygenation technique during intravenous deep sedation in pediatric dental treatment. The study is to evaluate the efficacy and safety of high-flow nasal oxygenation in intravenous deep sedation in pediatric dental patients.

ELIGIBILITY:
Inclusion Criteria:

1. children in need of deep sedation for dental treatment aged 3-7 years.
2. anticipated operation time over 60 mins.

Exclusion Criteria:

1. Conditions which the attending considers to be unfit for elective surgery or tubeless anesthesia.
2. Any contraindications of high flow nasal oxygenation.
3. Any contraindications or allergic history of propofol.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypoxemia | Intra-operative
  The occurrence of decreased oxygen saturation up to 90%.

SECONDARY OUTCOMES:
Severe Hypoxemia | Intra-operative
  The occurrence of decreased oxygen saturation up to 85%
Desaturation | Intra-operative
  The occurrence of decreased oxygen saturation up to 94%.
Intra-operative airway assistance | Intra-operative
  The need of intra-operative airway assistance maneuvers including jaw lifting, suction, mask ventilation and intubation.
Operation interruption | Intra-operative
  The occurrence of intra-operative surgical operation interruption due to decreased oxygen saturation, secretion, airway suction, severe body movement, etc., except for surgical reasons.
Intra-operative end-tidal carbon dioxide level | Intra-operative
  The highest intra-operative end-tidal carbon dioxide level.
Intra-operative transcutaneous carbon dioxide level | Intra-operative
  The highest intra-operative transcutaneous carbon dioxide level.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University of Stomatology, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided